CLINICAL TRIAL: NCT06016023
Title: Evaluation of Macrophage Inflammatory Protein-1α as a Periodontal Disease Biomarker in Oral Rinse: A Cross Sectional Study
Brief Title: Evaluation of Macrophage Inflammatory Protein-1α as a Periodontal Disease Biomarker
Status: Completed | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: RINDAPERIO2023
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis Chronic Generalized Severe; Gingivitis; Inflammatory Response
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: 30 periodontally healthy individuals.: Group 1 comprises of 30 periodontally healthy individuals who have never been clinically diagnosed with periodontitis.
- Group 2: 30 individuals with generalized gingivitis: Group 2 comprises of 30 participants diagnosed with generalized gingivitis according to the WWP 2017 classification.
- Group 3: 30 participants with generalised mild/moderate (STAGE I/II) periodontitis: Group 3 comprises of 30 participants, diagnosed with generalized mild/moderate (STAGE I/II) periodontitis, according to the WWP 2017 classification of periodontal disease.
- Group 4: 30 participants with generalized severe/very severe (STAGE III/IV) periodontitis: Group 4 comprises of 30 participants, diagnosed with generalized severe/very severe (STAGE III/IV) periodontitis, according to WWP 2017 classification of periodontal disease.

SUMMARY:
Periodontal disease is a chronic progressive state of inflammation pertaining to supporting tissues of the dentition that culminates in loss of the affected teeth. Currently, diagnosis and monitoring of periodontal disease progression is accomplished by performing a full-mouth clinical and radiological examination which is time-consuming and also requires elaborate infrastructure and equipment, which are not always available. Limitations of the conventional diagnostic techniques necessitate the development of point-of-care testing (POCT) which could serve as a rapid, feasible and affordable screening tool for periodontal disease.MIP-1α is a cysteine-cysteine (C-C) chemokine that is secreted by a variety of cells like macrophages, fibroblasts, epithelial cells and endothelial cells. They principally serve to recruit leukocytes like monocytes, T lymphocytes, natural killer cells, dendritic cells and granulocytes to the site of inflammation. Hence, the current study has a two fold aim; first, to determine the feasibility of MIP-1α as a periodontal disease biomarker; and second, to correlate the value of MIP-1α obtained from oral rinse sample with the periodontal disease severity.

DETAILED DESCRIPTION:
Periodontal disease is a chronic progressive state of inflammation pertaining to supporting tissues of the dentition that culminates in loss of the affected teeth. The term broadly covers both gingivitis (inflammation of the gingival connective tissue) and periodontitis (loss of supporting alveolar bone as a consequence of sustained inflammatory load on the supportive periodontal tissues). Currently, diagnosis and monitoring of periodontal disease progression is accomplished by performing a full-mouth clinical and radiological examination which is time-consuming and also requires elaborate infrastructure and equipment, which are not always available. These limitations of the conventional diagnostic techniques necessitate the development of point-of-care testing (POCT) which could serve as a rapid, feasible and affordable screening tool for periodontal disease.

Of late, chemokines have become the subject of interest for potential application as biomarkers for periodontal screening. MIP-1α is a cysteine-cysteine (C-C) chemokine that is secreted by a variety of cells like macrophages, fibroblasts, epithelial cells and endothelial cells. They principally serve to recruit leukocytes like monocytes, T lymphocytes, natural killer cells, dendritic cells and granulocytes to the site of inflammation. The primary challenge faced by researchers in analysis of host derived oral biomarkers in any sample fluid is the establishment of normal level of various biomarkers. This problem arises as the biomarkers that are found at exaggerated levels in periodontal inflammation are also detected in oral fluids in healthy periodontium but at a much lower value.

Hence, the current study has a two fold aim; first, to determine the feasibility of MIP-1α as a periodontal disease biomarker; and second, to correlate the value of MIP-1α obtained from oral rinse sample with the periodontal disease severity.

ELIGIBILITY:
Inclusion Criteria: Presence of ≥ 20 natural teeth

* Ability and willingness to give written informed consent
* Patients belonging to 4 groups -periodontally healthy, generalized gingivitis, generalized stage I/II periodontitis, generalized stage III/IV periodontitis

Exclusion Criteria:

* • Patients with chronic inflammatory disease such as nephrotic syndrome, chronic renal failure, significant cardiovascular disease, established type 1 or type 2 diabetes mellitus, or active cancer within the past 5 years

  * Smokers and alcoholics
  * Pregnant females
  * Presence of xerostomia
  * Patients with oral lesions or other contact sensitivity
  * Patients suffering from autoimmune diseases such as Sjogren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis
  * Patients with acute or chronic use of medications that cause oral dryness
  * Patients undergoing radiotherapy
  * Patients with Grade C periodontitis
  * Having received professional periodontal treatment within the previous 12 months
  * Having received antibiotic medication 3 months prior to study
  * Periapical pathology or other oral inflammatory conditions
  * Cognitive disability (interfering with ability to give samples)

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include consecutive subjects referred to the Department of Periodontics, PGIDS, Rohtak. The patients will be screened according to the inclusion and exclusion criteria for eligibility to participate in the study.
  The participants will comprise of the following groups :-
  1. Group 1: comprising of periodontally healthy individuals.
  2. Group 2: comprising of individuals, diagnosed with generalized gingivitis
  3. Group 3: comprising of participants, diagnosed with generalized mild/moderate (STAGE I/II) periodontitis
  4. Group 4: comprising of participants, diagnosed with generalized severe/very severe (STAGE III/IV) periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Macrophage Inflammatory Protein-1α (MIP-1α) level | 12-14 months
  Evaluation of MIP-1α level in sample across 4 groups of systemically healthy individuals (periodontally healthy, generalized gingivitis, generalized stage I/II periodontitis, generalized stage III/IV periodontitis)
To correlate the MIP-1α levels with clinical periodontal parameters | 12-14 months
  To correlate the MIP-1α levels with clinical periodontal parameters (Gingival Index, Clinical Attachment Loss, Bleeding On Probing, Probing Pocket Depth)

CONTACTS AND LOCATIONS:
Overall Officials: RINDA SHARMA, BDS, Principal Investigator — PT. B. D. SHARMA UHSR HARYANA
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India